CLINICAL TRIAL: NCT02740140
Title: Epidemiology of H. Pylori Transmission and Immunoepidemiology of Concomitant Infections
Brief Title: Epidemiology of H. Pylori Transmission
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: Santa Clara Valley Health & Hospital System (Other)
Responsible Party: Principal Investigator, Julie Parsonnet, Professor, Stanford University
Other Study IDs: SU-10182007-743
Record Dates: First submitted 2011-09-01; First posted 2016-04-15 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Communicable Diseases
Keywords: chronic coinfection
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum and PBMC
Oversight: Data Monitoring Committee: No

SUMMARY:
This observational epidemiologic study with nested cross-sectional and longitudinal aims will evaluate host immune response to mixed chronic infections (Helicobacter pylori, latent tuberculosis, intestinal helminthiasis) in recent US immigrants.

DETAILED DESCRIPTION:
1750 clinically-well, adult (age 18-55 years), recent immigrants (<2 years U.S. residence), referred through cooperating public health clinics in the Santa Clara Valley area, CA will be screened for H. pylori, helminth, and latent tuberculosis infections ["Screening" population]. Of these 1750, 426 will be selected for more intensive study (Cohort population), 105 of whom will receive baseline endoscopy. Of those selected for the cohort, 300 are expected to complete a 9-month follow-up assessment, 75 of whom are expected to undergo a second follow-up endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Between 18-55 years of age
* Either sex
* If female not pregnant or breastfeeding
* Lived in the United States less than 2 years
* Healthy
* Scheduled for Tuberculosis Skin Test (TST)

Exclusion Criteria:

* Under 18 and older than 55 years of age,
* Pregnant or breastfeeding
* Have lived in Unites States more that 2 years
* Chronic illness
* Not planning to get a TST

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 1750 clinically-well, adult (age 18-55 years), recent immigrants (<2 years U.S. residence), referred through cooperating public health clinics in the Santa Clara Valley area, CA will be screened for H. pylori, helminth, and latent tuberculosis infections ["Screening" population]. Of these 1750, 426 will be selected for more intensive study (Cohort population), 105 of whom will receive baseline endoscopy. Of those selected for the cohort, 300 are expected to complete a 9-month follow-up assessment, 75 of whom are expected to undergo a second follow-up endoscopy.
Sampling Method: Non-Probability Sample
Enrollment: 1750 (Actual)
Dates: Start 2008-06; Primary Completion 2011-06 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Change in cytokine responses from baseline at 9 months in TB and H. pylori antigen-induced PBMC before and after provider managed treatment of latent TB or helminth infection | Baseline and 9 months after treatment for either latent TB or helminth infections; analyzed after all subjects recruited (3 years of recruitment plus 9 months follow-up).

SECONDARY OUTCOMES:
Correlation of cytokine response to TB antigens and helminths with humoral responses to infections with H. pylori. | Assays performed when collected over three years from recruited subjects; analyzed at the end of three years.
Population prevalence of individual and joint infections with H pylori, latent tuberculosis, heminthiasis in recent immigrant to northern California | Assays performed when collected over three years from recruited subjects; analyzed at the end of three years.
  We compare prevalence of these infections in recent immigrants by geographic area

CONTACTS AND LOCATIONS:
Overall Officials: Julie Parsonnet, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Santa Clara Public Health Clinics, San Jose, California
  - Stanford University School of Medicine, Stanford, California

REFERENCES:
- [Background] Chang AH, Perry S, Du JN, Agunbiade A, Polesky A, Parsonnet J. Decreasing intestinal parasites in recent Northern California refugees. Am J Trop Med Hyg. 2013 Jan;88(1):191-7. doi: 10.4269/ajtmh.2012.12-0349. Epub 2012 Nov 13. PMID 23149583
- [Background] Perry S, Chang AH, Sanchez L, Yang S, Haggerty TD, Parsonnet J. The immune response to tuberculosis infection in the setting of Helicobacter pylori and helminth infections. Epidemiol Infect. 2013 Jun;141(6):1232-43. doi: 10.1017/S0950268812001823. Epub 2012 Sep 7. PMID 22954328
- [Background] Herrera V, Perry S, Parsonnet J, Banaei N. Clinical application and limitations of interferon-gamma release assays for the diagnosis of latent tuberculosis infection. Clin Infect Dis. 2011 Apr 15;52(8):1031-7. doi: 10.1093/cid/cir068. PMID 21460320
- [Background] Perry S, Hussain R, Parsonnet J. The impact of mucosal infections on acquisition and progression of tuberculosis. Mucosal Immunol. 2011 May;4(3):246-51. doi: 10.1038/mi.2011.11. Epub 2011 Mar 16. PMID 21412228